CLINICAL TRIAL: NCT03055936
Title: A Dose-finding Study for Levodopa, Carbidopa and ODM-104 Test Formulations After Repeated Administration in Healthy Males
Brief Title: Dose-finding Pharmacokinetic Study in Healthy Males
Acronym: COMDOS1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3112005
Record Dates: First submitted 2017-01-20; First posted 2017-02-16 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Levodopa; carbidopa, levodopa drug combination; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- A1 (Experimental): levodopa 50 mg, carbidopa 12.5 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- B1 (Experimental): levodopa 50 mg, carbidopa 65 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- C1 (Experimental): levodopa 50 mg, carbidopa 65 mg, ODM-104 50 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- D1 (Experimental): levodopa 50 mg, carbidopa 65 mg, ODM-104 100 mg A4 ; B4 l; C4 ; D4 levodopa 100 mg, carbidopa 65 mg, ODM-104 100 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- A2 (Experimental): levodopa 100 mg, carbidopa 25 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- B2 (Experimental): levodopa 100 mg, carbidopa 65 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- C2 (Experimental): levodopa 100 mg, carbidopa 65 mg, ODM-104 50 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- D2 (Experimental): levodopa 100 mg, carbidopa 37,5 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- A3 (Experimental): levodopa 150 mg, carbidopa 65 mg, ODM-104 100 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- B3 (Experimental): levodopa 150 mg, carbidopa 65 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- C3 (Experimental): levodopa 150 mg, carbidopa 65 mg, ODM-104 50 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- D3 (Experimental): levodopa 150 mg, carbidopa 65 mg, ODM-104 100 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- A4 (Experimental): levodopa IR 100 mg (Sinemet), carbidopa 25 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- B4 (Experimental): levodopa 100 mg, carbidopa 65 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa
- C4 (Experimental): levodopa 100 mg, carbidopa 25 mg, ODM-104 100 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104
- D4 (Experimental): levodopa 100 mg, carbidopa 65 mg, ODM-104 100 mg
  Interventions: Drug: Levodopa; Drug: Carbidopa; Drug: ODM-104

INTERVENTIONS:
Drug: Levodopa — Levodopa 50 mg or 100 mg or 150 mg
  Other Names: Sinemet
Drug: Carbidopa — Carbidopa 12.5 mg or 25 mg or 65 mg
Drug: ODM-104 — ODM-104 50 mg or 100 mg
  Arms: A3; C1; C2; C3; C4; D1; D3; D4

SUMMARY:
This is a phase I PK study in healthy males.

DETAILED DESCRIPTION:
This is a phase I, open, repeated dose, randomised PK study in healthy males. The study will consist of 4 parallel groups (Groups 1-4). All groups will have a crossover design with 4 treatment periods, each lasting for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history and physical examinations.
* Males between 18-65 years of age inclusive at screening.
* Body mass index (BMI) between 19-30 kg/m2 (BMI = weight/height2) inclusive at screening.
* Weight at least 55 kg inclusive at screening.
* Regular intestinal transit (no recent history of recurrent constipation, diarrhoea, or other intestinal problems, and no history of major gastrointestinal surgery).
* Subject with a partner of childbearing potential agrees to use adequate contraception from the first dose of study treatment until 90 days after the last dose of study treatment. Adequate methods of contraception include: Hormonal contraceptives, barrier methods (condom, diaphragm, cervical cap, etc.) in combination with a spermicide, intrauterine device and sexual abstinence.
* Subject agrees to not donate sperm from the first dose of study treatment until 90 days after the last dose of study treatment.

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic, endocrine, neurological or psychiatric disease or cancer (except local non-melanoma skin cancer) within the previous 2 years.
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, paracetamol for occasional pain is allowed.
* Any clinically significant abnormal laboratory value or ECG (such as prolonged QTcF >450 ms or QRS >120 ms) that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject if he takes part in the study.
* Known hypersensitivity to the active substances or the excipients of the drugs.
* History of vasovagal collapses or vagal reactions with unexplained reason within the previous 2 years or a tendency for vasovagal reactions during blood sampling.
* HR < 50 bpm or > 90 bpm in the supine position after 5 min rest at the screening visit.
* At the screening visit:

  * systolic BP < 100 mmHg or > 140 mmHg in the supine position after 5 min rest
  * diastolic BP < 50 mmHg or > 90 mmHg in the supine position after 5 min rest.
* Creatinine > 1.5 x upper limit of normal (ULN) and alanine aminotransferase or aspartate aminotransferase >1.25 x ULN at screening.
* History of anaphylactic/anaphylactoid reactions.
* Strong tendency to motion sickness.
* Recent or current (suspected) drug abuse.
* Recent or current alcohol abuse; regular drinking of more than 21 units per week (1 unit = 4 cl spirits or equivalent).
* Current use of nicotine-containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine-containing products for 48 h before the first dose in each period until collection of the 24 h PK sample in the morning of day 8.
* Use of caffeine-containing beverages more than 600 mg of caffeine/day and/or inability to refrain from using caffeine-containing beverages 24 h before the first levodopa administration on the PK day (day 7) until collection of the 24 h PK sample in the morning of day 8.
* Blood donation or loss of a significant amount of blood (> 500 ml) within 90 days before the first study treatment administration.
* Participation in another investigational drug study or administration of another investigational drug within 60 days before the first study treatment administration.
* Veins unsuitable for repeated venipuncture or cannulation.
* Predictable poor compliance or inability to communicate well with the study centre personnel.
* Inability to participate in all treatment periods.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Strugala, DR.med., Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan Pharma Services, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: A1 levodopa 50 mg, carbidopa 12.5 mg; B1 levodopa 50 mg, carbidopa 65 mg; C1 levodopa 50 mg, carbidopa 65 mg, ODM-104 50 mg; D1 levodopa 50 mg, carbidopa 65 mg, ODM-104 100 mg
- Group 2: A2 levodopa 100 mg, carbidopa 25 mg; B2 levodopa 100 mg, carbidopa 65 mg; C2 levodopa 100 mg, carbidopa 65 mg, ODM-104 50 mg; D2 levodopa 100 mg, carbidopa 65 mg, ODM-104 100 mg
- Group 3: A3 levodopa 150 mg, carbidopa 37.5 mg; B3 levodopa 150 mg, carbidopa 65 mg; C3 levodopa 150 mg, carbidopa 65 mg, ODM-104 50 mg; D3 levodopa 150 mg, carbidopa 65 mg, ODM-104 100 mg
- Group 4: A4 (Sinemet: levodopa IR 100 mg, carbidopa 25 mg; B4 levodopa 100 mg, carbidopa 65 mg; C4 levodopa 100 mg, carbidopa 25 mg, ODM-104 100 mg; D4 levodopa 100 mg, carbidopa 65 mg, ODM-104 100 mg
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 14 | 14 | 14 | 14
Completed | 12 | 13 | 12 | 13
Not Completed | 2 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Personal reason | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 4: A4 (Sinemet): levodopa IR 100 mg, carbidopa 25 mg; B4 levodopa 100 mg, carbidopa 65 mg; C4 levodopa 100 mg, carbidopa 25 mg, ODM-104 100 mg; D4 levodopa 100 mg, carbidopa 65 mg, ODM-104 100 mg
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 14 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — The figures given per group are per performed statistical analysis.
  years | 42.4 (13.7) | 49.5 (10.9) | 48.0 (13.5) | 46.0 (10.6) | 46.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 14 | 14 | 14 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 14 | 14 | 14 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 13 | 13 | 13 | 13 | 52
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 14 | 14 | 14 | 14 | 14

OUTCOME MEASURES:

1. Primary Outcome: Levodopa Area Under the Concentration-time Curve From Time 0 to the 24 h PK Sample (AUC0-24) Time 0 to the 24 h PK Sample (AUC0-24)
Description: Levodopa Area Under the Concentration-time Curve From Time 0 to the 24 h PK Sample (AUC0-24)
Time Frame: During 24 hours
Population: PP (Per Protocol population)
Measure: Mean (90% Confidence Interval); unit: h*ng/ml
Groups:
- A1 50 mg LD + 12.5 mg CD: 50 mg of MR levodopa + 12.5 mg of carbidopa
- B1 50 mg LD + 65 mg CD: 50 mg of MR levodopa + 65 mg of carbidopa
- C1 50 mg LD + 65 mg CD + 50 mg ODM-104: 50 mg of MR levodopa + 65 mg carbidopa + 50 mg ODM-104
- D1 50 mg LD + 65 mg CD + 100 mg ODM-104: 50 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104
- A2 100 mg LD + 25 mg CD: 100 mg of MR levodopa + 25 mg of carbidopa
- B2 100 mg LD + 65 mg CD; B4 100 mg LD + 65 mg CD: 100 mg of MR levodopa + 65 mg of carbidopa
- C2 100 mg of LD + 65 mg CD + 50 mg ODM-104: 100 mg of MR levodopa + 65 mg of carbidopa + 50 mg of ODM-104
- D2 100 mg LD + 65 mg CD + 100 mg of ODM-104; D4 100 mg LD + 65 mg CD + 100 mg ODM-104: 100 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104
- A3 150 mg LD + 37.5 mg CD: 150 mg of MR levodopa + 37.5 mg of carbidopa
- B3 150 mg LD + 65 mg CD: 150 mg of MR levodopa + 65 mg of carbidopa
- C3 150 mg LD + 65 mg CD + 50 mg ODM-104: 150 mg of MR levodopa + 65 mg of carbidopa + 50 mg of ODM-104
- D3 150 mg LD + 65 mg CD + 100 mg ODM-104: 150 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104
- A4 (Sinemet) 100 mg IR LD + 25 mg CD: (Sinemet) 100 mg of IR levodopa + 25 mg of carbidopa
- C4 100 mg LD + 25 mg CD + 100 mg ODM-104: 100 mg of MR levodopa + 25 mg of carbidopa + 100 mg of ODM-104
Arm/Group | A1 50 mg LD + 12.5 mg CD | B1 50 mg LD + 65 mg CD | C1 50 mg LD + 65 mg CD + 50 mg ODM-104 | D1 50 mg LD + 65 mg CD + 100 mg ODM-104 | A2 100 mg LD + 25 mg CD | B2 100 mg LD + 65 mg CD | C2 100 mg of LD + 65 mg CD + 50 mg ODM-104 | D2 100 mg LD + 65 mg CD + 100 mg of ODM-104 | A3 150 mg LD + 37.5 mg CD | B3 150 mg LD + 65 mg CD | C3 150 mg LD + 65 mg CD + 50 mg ODM-104 | D3 150 mg LD + 65 mg CD + 100 mg ODM-104 | A4 (Sinemet) 100 mg IR LD + 25 mg CD | B4 100 mg LD + 65 mg CD | C4 100 mg LD + 25 mg CD + 100 mg ODM-104 | D4 100 mg LD + 65 mg CD + 100 mg ODM-104
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 13 | 13 | 13 | 13 | 12 | 12 | 12 | 12 | 13 | 13 | 13 | 13
h*ng/ml | 4300 [3905 to 4734] | 5423 [4928 to 5968] | 7439 [6760 to 8186] | 9046 [8215 to 9960] | 9643 [9060 to 10263] | 10709 [10062 to 11399] | 15257 [14335 to 16239] | 17896 [16814 to 19048] | 14285 [13550 to 15061] | 15805 [14995 to 16658] | 22473 [21316 to 23693] | 25672 [24390 to 27021] | 7965 [6436 to 9859] | 8994 [7286 to 11104] | 13866 [11232 to 17118] | 16310 [13140 to 20246]

2. Secondary Outcome: Fluctuation of Levodopa Cmax/Cmin, Tau
Description: Explore fluctuation of levodopa Cmax/Cmin, tau. Figures given are per performed statistical analysis.
Time Frame: 16 hours
Measure: Mean (Standard Deviation); unit: (ng/ml)/(ng/ml)
Arm/Group | A1 50 mg LD + 12.5 mg CD | B1 50 mg LD + 65 mg CD | C1 50 mg LD + 65 mg CD + 50 mg ODM-104 | D1 50 mg LD + 65 mg CD + 100 mg ODM-104 | A2 100 mg LD + 25 mg CD | B2 100 mg LD + 65 mg CD | C2 100 mg of LD + 65 mg CD + 50 mg ODM-104 | D2 100 mg LD + 65 mg CD + 100 mg of ODM-104 | A3 150 mg LD + 37.5 mg CD | B3 150 mg LD + 65 mg CD | C3 150 mg LD + 65 mg CD + 50 mg ODM-104 | D3 150 mg LD + 65 mg CD + 100 mg ODM-104 | A4 (Sinemet) 100 mg IR LD + 25 mg CD | B4 100 mg LD + 65 mg CD | C4 100 mg LD + 25 mg CD + 100 mg ODM-104 | D4 100 mg LD + 65 mg CD + 100 mg ODM-104
Number analyzed (Participants) | 13 | 14 | 14 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 14 | 14 | 13
(ng/ml)/(ng/ml) | 12.24 (5.73) | 7.49 (2.23) | 4.16 (0.77) | 3.02 (1.00) | 11.00 (3.30) | 8.32 (2.23) | 4.46 (1.09) | 3.35 (0.74) | 8.45 (3.16) | 7.16 (3.87) | 3.67 (1.29) | 2.82 (0.99) | 19.52 (14.13) | 9.18 (6.23) | 7.63 (12.96) | 3.04 (0.76)

3. Secondary Outcome: Levodopa Peak Plasma Concentration (Cmax)
Description: Levodopa peak plasma concentration (Cmax)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | A1 50 mg LD + 12.5 mg CD | B1 50 mg LD + 65 mg CD | C1 50 mg LD + 65 mg CD + 50 mg ODM-104 | D1 50 mg LD + 65 mg CD + 100 mg ODM-104 | A2 100 mg LD + 25 mg CD | B2 100 mg LD + 65 mg CD | C2 100 mg of LD + 65 mg CD + 50 mg ODM-104 | D2 100 mg LD + 65 mg CD + 100 mg of ODM-104 | A3 150 mg LD + 37.5 mg CD | B3 150 mg LD + 65 mg CD | C3 150 mg LD + 65 mg CD + 50 mg ODM-104 | D3 150 mg LD + 65 mg CD + 100 mg ODM-104 | A4 (Sinemet) 100 mg IR LD + 25 mg CD | B4 100 mg LD + 65 mg CD | C4 100 mg LD + 25 mg CD + 100 mg ODM-104 | D4 100 mg LD + 65 mg CD + 100 mg ODM-104
Number analyzed (Participants) | 13 | 14 | 14 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 14 | 14 | 13
ng/ml | 685.92 (193.08) | 775.36 (186.29) | 908.86 (230.23) | 950.38 (241.60) | 1519.92 (294.51) | 1593.85 (288.95) | 1855.38 (240.58) | 1955.38 (278.62) | 2105.45 (422.05) | 2072.73 (403.78) | 2545.45 (424.30) | 2616.67 (388.76) | 1634.62 (361.70) | 1367.36 (352.26) | 1711.43 (316.10) | 1717.69 (641.60)

ADVERSE EVENTS:
Time Frame: Through study completion, upto 15 weeks.
Description: Adverse events are recorded per arm. Same applies to Number of Participants at Risk across the All-Cause Mortality, Serious Adverse Events and/or Other (Not Including Serious) Adverse Events.
Groups:
- A1 (Levodopa 50, Carbidopa 12.5): levodopa 50 mg, carbidopa 12.5 mg
- B1 (Levodopa 50, Carbidopa 65): levodopa 50 mg, carbidopa 65 mg
- C1 (Levodopa 50, Carbidopa 65, ODM-104 50): levodopa 50 mg, carbidopa 65 mg, ODM-104 50 mg
- D1 (Levodopa 50, Carbidopa 65, ODM-104 100): levodopa 50 mg, carbidopa 65 mg, ODM-104 100 mg
- A2 (levodopa100, Carbidopa 25): levodopa 100 mg, carbidopa 25 mg
- B2 (Levodopa 100, Carbidopa 65); B4 (Levodopa 100, Carbidopa 65): levodopa 100 mg, carbidopa 65 mg
- C2 (levodopa100, Carbidopa 65, ODM-104 50): levodopa 100 mg, carbidopa 65 mg, ODM-104 50 mg
- D2 (Levodopa 100, Carbidopa 65, ODM-104 100); D4 (Levodopa 100, Carbidopa 65, ODM-104 100): levodopa 100 mg, carbidopa 65 mg, ODM-104 100 mg
- A3 (Levodopa 150, Carbidopa 37.5): levodopa 150 mg, carbidopa 37.5 mg;
- B3 (Levodopa 150, Carbidopa 65): levodopa 150 mg, carbidopa 65 mg
- C3 (Levodopa 150, Carbidopa 65, ODM-104 50): levodopa 150 mg, carbidopa 65 mg, ODM-104 50 mg
- D3 (Levodopa 150, Carbidopa 65, ODM-104 100): levodopa 150 mg, carbidopa 65 mg, ODM-104 100 mg
- A4 (Sinemet, Levodopa 100, Carbidopa 25): levodopa IR (Sinemet) 100 mg, carbidopa 25 mg
- C4 (Levodopa 100, Carbidopa 25, ODM-104 100): levodopa 100 mg, carbidopa 25 mg, ODM-104 100 mg
Arm/Group | A1 (Levodopa 50, Carbidopa 12.5) | B1 (Levodopa 50, Carbidopa 65) | C1 (Levodopa 50, Carbidopa 65, ODM-104 50) | D1 (Levodopa 50, Carbidopa 65, ODM-104 100) | A2 (levodopa100, Carbidopa 25) | B2 (Levodopa 100, Carbidopa 65) | C2 (levodopa100, Carbidopa 65, ODM-104 50) | D2 (Levodopa 100, Carbidopa 65, ODM-104 100) | A3 (Levodopa 150, Carbidopa 37.5) | B3 (Levodopa 150, Carbidopa 65) | C3 (Levodopa 150, Carbidopa 65, ODM-104 50) | D3 (Levodopa 150, Carbidopa 65, ODM-104 100) | A4 (Sinemet, Levodopa 100, Carbidopa 25) | B4 (Levodopa 100, Carbidopa 65) | C4 (Levodopa 100, Carbidopa 25, ODM-104 100) | D4 (Levodopa 100, Carbidopa 65, ODM-104 100)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 2/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 6/14 | 8/14 | 7/14 | 7/14 | 6/14 | 7/14 | 8/14 | 7/14 | 7/14 | 4/14 | 9/14 | 10/14 | 6/14 | 5/14 | 5/14 | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 (Levodopa 50, Carbidopa 12.5) (N=14) | B1 (Levodopa 50, Carbidopa 65) (N=14) | C1 (Levodopa 50, Carbidopa 65, ODM-104 50) (N=14) | D1 (Levodopa 50, Carbidopa 65, ODM-104 100) (N=14) | A2 (levodopa100, Carbidopa 25) (N=14) | B2 (Levodopa 100, Carbidopa 65) (N=14) | C2 (levodopa100, Carbidopa 65, ODM-104 50) (N=14) | D2 (Levodopa 100, Carbidopa 65, ODM-104 100) (N=14) | A3 (Levodopa 150, Carbidopa 37.5) (N=14) | B3 (Levodopa 150, Carbidopa 65) (N=14) | C3 (Levodopa 150, Carbidopa 65, ODM-104 50) (N=14) | D3 (Levodopa 150, Carbidopa 65, ODM-104 100) (N=14) | A4 (Sinemet, Levodopa 100, Carbidopa 25) (N=14) | B4 (Levodopa 100, Carbidopa 65) (N=14) | C4 (Levodopa 100, Carbidopa 25, ODM-104 100) (N=14) | D4 (Levodopa 100, Carbidopa 65, ODM-104 100) (N=14)
Diverticulitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 (Levodopa 50, Carbidopa 12.5) (N=14) | B1 (Levodopa 50, Carbidopa 65) (N=14) | C1 (Levodopa 50, Carbidopa 65, ODM-104 50) (N=14) | D1 (Levodopa 50, Carbidopa 65, ODM-104 100) (N=14) | A2 (levodopa100, Carbidopa 25) (N=14) | B2 (Levodopa 100, Carbidopa 65) (N=14) | C2 (levodopa100, Carbidopa 65, ODM-104 50) (N=14) | D2 (Levodopa 100, Carbidopa 65, ODM-104 100) (N=14) | A3 (Levodopa 150, Carbidopa 37.5) (N=14) | B3 (Levodopa 150, Carbidopa 65) (N=14) | C3 (Levodopa 150, Carbidopa 65, ODM-104 50) (N=14) | D3 (Levodopa 150, Carbidopa 65, ODM-104 100) (N=14) | A4 (Sinemet, Levodopa 100, Carbidopa 25) (N=14) | B4 (Levodopa 100, Carbidopa 65) (N=14) | C4 (Levodopa 100, Carbidopa 25, ODM-104 100) (N=14) | D4 (Levodopa 100, Carbidopa 65, ODM-104 100) (N=14)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 3 (5) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 4 (5) | 4 (8) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 4 (10) | 1 (1) | 3 (9)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 1 (2) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (7) | 1 (1) | 1 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decrease appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site dryness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03055936/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03055936/SAP_001.pdf